CLINICAL TRIAL: NCT00958854
Title: Phase II Trial of Fludarabine & Cyclophosphamide Followed by Thalidomide for Angioimmunoblastic Lymphoma
Brief Title: Fludarabine, Cyclophosphamide, and Thalidomide in Treating Patients With Angioimmunoblastic T-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000644123; CRUK-UCL-AITL; EUDRACT-2005-003931-40; EU-20947
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Lymphoma
Keywords: angioimmunoblastic T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Immunoblastic Lymphadenopathy | interventions — Cyclophosphamide; fludarabine phosphate; Thalidomide

INTERVENTIONS:
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: thalidomide
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Thalidomide may stop the growth of lymphoma by blocking blood flow to the cancer. Giving fludarabine and cyclophosphamide together with thalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving fludarabine and cyclophosphamide together with thalidomide works in treating patients with angioimmunoblastic T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with angioimmunoblastic T-cell lymphoma after chemotherapy comprising fludarabine and cyclophosphamide.

Secondary

* Assess the incremental anatomical and molecular response rate in these patients during treatment with thalidomide.
* Determine the toxicity of treatment with fludarabine and cyclophosphamide followed by thalidomide.
* Assess the progression-free and overall survival of these patients.
* Develop a detailed pathological description of the disease at presentation and at relapse.
* Assess the number of circulating clonal T cells at presentation and during thalidomide treatment.
* Screen for possible etiological viruses at presentation.
* Evaluate the evolution of EBV viral load during follow-up.

OUTLINE: This is a multicenter study.

Patients receive oral or IV fludarabine and oral or IV cyclophosphamide once daily on days 1-3. Courses repeat every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity. Beginning at least 4 weeks after completion of chemotherapy, patients who achieve at least stable disease receive oral thalidomide once daily for at least 6 months.

Lymph nodes, marrow, and peripheral blood will be collected periodically for research studies.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed angioimmunoblastic T-cell lymphoma
* Measurable disease (i.e., anatomically assessable)

PATIENT CHARACTERISTICS:

* WHO/ECOG performance status 0-2
* Serum creatinine ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and after study treatment
* No known seropositivity for hepatitis B virus, hepatitis C virus, or HIV
* No active second malignancy or other concomitant serious medical condition, in particular peripheral neuropathy

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for angioimmunoblastic T-cell lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2006-01; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Response rate after chemotherapy with fludarabine and cyclophosphamide

SECONDARY OUTCOMES:
Incremental response rate to thalidomide treatment
Toxicity according to the NCI CTCAE v.3.0
Progression-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Claudius Rudin, MD, Principal Investigator — Royal Devon and Exeter Hospital
Locations (1):
- Cancer Research UK and University College London Cancer Trials Centre, Exeter, England, United Kingdom